CLINICAL TRIAL: NCT02226536
Title: Fractionated and Restrictive Glucose Diet in Patients With Vestibular Dysfunction: a Randomized Controlled Trial
Brief Title: Vestibular Dysfunction and Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Roseli Saraiva Moreira Bittar, Assistente Doutor da Faculdade de Medicina da Universidade de São Paulo, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMG-PDCEAV
Record Dates: First submitted 2014-08-06; First posted 2014-08-27 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Dysfunction of Vestibular System; Glucose Intolerance
Keywords: Posture; Vertigo; glucose metabolism; diet; scales; dinamic posturography
MeSH Terms: conditions — Glucose Intolerance; Vertigo | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): Usual diet without any orientation
  Interventions: Behavioral: fractioned diet without glucose
- fractioned diet without glucose (Active Comparator): Fractioned diet without glucose
  Interventions: Behavioral: fractioned diet without glucose

INTERVENTIONS:
Behavioral: fractioned diet without glucose — Patients were divided into two groups: Diet Group was treated with placebo pills and glucose restrictive and fractionated diet. Control Group received only placebo pills. All individuals had their vestibular function evaluated by Computerized Dynamic Posturography and done visual analogue scale (VAS) in the first day and 30 days after diet intervention

SUMMARY:
Introduction: the global sugar consumption has increased in the past 50 years and their abusive intake is responsible for the insulin resistance and causes the metabolic syndrome - obesity, diabetes mellitus, hypertension and coronary heart disease. Objective: To evaluate the effect of scheduled diet without glucose as treatment of labyrinthine disorders associated with glucose-insulin index. Study Design: A prospective randomized controlled trial. Patients and Methods: A study conducted at the University of São Paulo with 51 patients divided into two groups: Diet Group (DG) that comprises subjects treated with fractionated diet with glucose restriction and control group (CG) where individuals were not counseled regarding diet. Patients underwent computerized dynamic posturography - sensory organization test (CDP - SOT) and Visual Analog Scale (VAS) in the first and thirtieth days of the study.

DETAILED DESCRIPTION:
51 patientes with dizziness and glucose intolerance diagnosed by the glucose tolerance test were selected.

The subjects were submited to CDP SOT conditions and a visual analogue scale to measure his self perception about dizziness.

Then, they were randomized in two groups: with and without fractioned diet without glucose during 30 days.

The CDP was repeated in order to verify a statistical difference of SOT condition 5 that reflects the individual hability to maintain the own posture with the vestibule solely and CS - that represents the final balance situation.

The VAS was repeated too in order to verify the self perception of the dizziness after diet.

ELIGIBILITY:
Inclusion Criteria:

* dizziness related to fasting or glucose intake
* alterations of glucose tolerance test

Exclusion Criteria:

* dizziness not related to vestibular problems
* ortopedical or neurological diseases
* diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assessment of equilibrium score through the computerized dynamic posturography (CDP) in 51 patients | 30 days

SECONDARY OUTCOMES:
Self perception of dizziness mesured by the visual analogue scale | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Roseli SM Bittar, MD, PhD, Principal Investigator — University of Sao Paulo